CLINICAL TRIAL: NCT01114230
Title: A Phase 1, Open-label, Multi-center, Dose Escalation Study of the Safety and Pharmacokinetics of AGS-16M8F Monotherapy in Subjects With Advanced Renal Cell Carcinoma
Brief Title: A First in Man Study to Determine the Safety at Various Dose Levels of AGS-16M8F in Advanced Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Agensys, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009002
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Renal Cell Carcinoma; Pharmacokinetics of AGS-16M8F
Keywords: Advanced Renal Cell Carcinoma; Advanced Kidney Cancer; AGS-16M8F
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Dose Level 1 (Experimental)
  Interventions: Drug: AGS-16M8F
- Dose Level 2 (Experimental)
  Interventions: Drug: AGS-16M8F
- Dose Level 3 (Experimental)
  Interventions: Drug: AGS-16M8F
- Dose Level 4 (Experimental)
  Interventions: Drug: AGS-16M8F
- Dose Level 5 (Experimental)
  Interventions: Drug: AGS-16M8F
- Dose Level 6 (Experimental)
  Interventions: Drug: AGS-16M8F
- Dose Level 7 (Experimental)
  Interventions: Drug: AGS-16M8F
- Dose Level 8 (Experimental)
  Interventions: Drug: AGS-16M8F
- Dose Level 9 (Experimental)
  Interventions: Drug: AGS-16M8F

INTERVENTIONS:
Drug: AGS-16M8F — IV

SUMMARY:
The purpose of this dose escalation study is to examine the safety and pharmacokinetics (PK) of AGS-16M8F administered in subjects with advanced renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis (recent or remote) of metastatic renal cell carcinoma (including papillary, clear cell, and excluding transitional cell types) that is not amenable to cure by surgery or other means.
* Non-measurable or measurable disease according to Response Criteria for Solid Tumors (RECIST Version 1.1)
* Eastern Cooperative Group (ECOG) performance status of 0-1
* Negative pregnancy test (women of childbearing potential)
* Hematologic function, as follows:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelet count ≥ 100 x 109/L
  * Hemoglobin ≥ 9 g/dL (transfusions are allowed)
* Renal function, as follows:

  * creatinine ≤ 1.5 x upper limit of normal (ULN), or calculated glomerular filtration rate (GFR) > 50 mL/min if creatinine > 1.5x ULN
* Hepatic function, as follows:

  * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 x ULN or ≤ 5x ULN if known liver metastases
  * Total bilirubin ≤ 1.5 x ULN
* International Normalized Ratio (INR) < 1.3 (or ≤ 3.0 if on therapeutic anticoagulation)
* Women and men of childbearing potential must be advised and agree to practice effective methods of contraception during the course of the study and for four weeks after the last AGS-16M8F infusion administration

Exclusion Criteria:

* Past or present documented central nervous system (CNS) tumor or CNS metastasis
* Use of any investigational drug (including marketed drugs not approved for this indication) within 4 weeks prior to screening
* History of thromboembolic events and bleeding disorders ≤ 3 months (e.g., DVT or PE)
* Active angina or Class III or IV Congestive Heart Failure (New York Heart Association CHF Functional Classification System) or clinically significant cardiac disease within 12 months of study enrollment, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, congestive heart failure, uncontrolled hypertension, or arrythmias not controlled by outpatient medication
* Major surgery (that requires general anesthesia) within 4 weeks of study enrollment
* Women who are pregnant (confirmed by positive pregnancy test) or lactating
* Known positive test for human immunodeficiency virus (HIV), hepatitis C, or hepatitis B surface antigen
* Active infection requiring treatment with systemic (intravenous or oral) anti-infectives (antibiotic, antifungal, or antiviral agent) within 72 hours of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety assessed by recording adverse events, vital signs and laboratory assessments | For 12 weeks during treatment period and up to 4 weeks follow up
Pharmacokinetic variables assessment through analysis of blood samples | Up to day 15 for cycle 1 and cycle 4 and pre-dose for cycles 2 and 3; every 3 weeks during the second 12 weeks of treatment; and if subject continues on study drug, every 12 weeks thereafter

SECONDARY OUTCOMES:
Incidence of anti-AGS-16M8F antibody formation | Baseline; up to day 64 during the first 12 weeks; and if subject continues on study drug, every 3 weeks during the second 12 weeks of treatment and every 12 weeks thereafter
Incidence of Tumor Response (complete or partial response) | Baseline and every 12 weeks while on study drug

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Agensys, Inc.
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Seattle Cancer Care Alliance, Seattle, Washington